CLINICAL TRIAL: NCT00876356
Title: Conjugated Linoleic Acid (CLA) as Adjunctive Therapy in Mild Asthmatics: A Pilot Study.
Brief Title: The Health Benefits of Conjugated Linoleic Acid (CLA) for Asthma & Allergy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Canadian Lung Association/British Columbia Lung Association (Unknown); Natural Inc./Cognis GmbH (Dusseldorf, Germany) (Unknown)
Responsible Party: Dr. Delbert R. Dorscheid, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P01-0180
Record Dates: First submitted 2009-04-03; First posted 2009-04-06 (Estimated); Last update posted 2009-04-06 (Estimated); Status verified 2009-04

CONDITIONS: Asthma
Keywords: Asthma; Conjugated Linoleic Acid (CLA); dietary supplement
MeSH Terms: conditions — Asthma | interventions — Linoleic Acids, Conjugated; Olive Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Conjugated Linoleic Acid 4.5g/day in three divided doses p.o. for 12 weeks
  Interventions: Dietary Supplement: Conjugated Linoleic Acid (CLA)
- 2 (Placebo Comparator): Olive oil 4.5g/day x 12 weeks.
  Interventions: Dietary Supplement: Olive oil

INTERVENTIONS:
Dietary Supplement: Conjugated Linoleic Acid (CLA) — CLA 4.5g/day in three divided doses p.o. for 12 weeks
  Arms: 1
Dietary Supplement: Olive oil — Olive oil 4.5g/day x 12 weeks
  Arms: 2

SUMMARY:
Conjugated linoleic acids (CLA) are naturally occurring free fatty acids derived from the tissues and milk of ruminant animals such as cows. CLA has multiple biological properties including regulation of metabolism and immune processes, including tissue inflammation. Asthma symptoms are caused by irritation and inflammation of the airways. Our hypothesis was that CLA may reduce airway inflammation in asthma and thus reduce asthma symptoms. The aim of this pilot study was to investigate the efficacy and safety of CLA as a dietary supplement in mild asthma. Subjects will be assigned to take CLA dietary supplements or placebo (olive oil) for 12 weeks in addition to their usual asthma treatment. They will be monitored for asthma symptoms, side effects, lung function and blood markers of inflammation.

DETAILED DESCRIPTION:
Background and Purpose You are being invited to participate in a study of the effects of a natural supplement, conjugated linoleic acid (CLA), on allergy and asthma. Previous studies show that CLA may control the type of inflammation found in allergy and asthma. CLA is found in dairy products, however the amount found varies greatly depending on what the cows have been fed and has reduced dramatically over the last 30 years. The estimated daily intake of CLA is between 15 and 174 mg/day, but an effective dose of CLA is 3000 to 4000 mg/day for a 70 kg adult. Therefore taking CLA supplements may be beneficial. This will be the first formal study to look at whether CLA does benefit people with allergies and asthma.

Study Procedures

If you qualify for the study and agree to participate, you will be randomly assigned (like flipping a coin) into one of two groups. The two groups are:

Conjugated linoleic acid (active substance) twice daily for 3 months Placebo (inactive substance) twice daily for 3 months

Neither you nor the study doctors will know whether you are receiving CLA or placebo. There will be no change in your asthma medications that are prescribed by your regular physician. Your physician will be made aware that you are participating in this study.

Your participation in the study involves 6 visits to our laboratory, of about 2 hours duration each. The study will run for 3 months.

At 4 of the visits, which will happen every 4 weeks, you will be asked to perform spirometry and sputum induction. Spirometry is a breathing test which requires you to take a deep breath in and blow it out as hard and fast as you can. From this we can measure baseline airway function. This takes about 15 minutes, has no side effects and is a routinely performed test on patients in our clinical pulmonary function laboratory.

Sputum induction involves the inhalation of a mist of salt water to help produce a deep cough and a sputum sample from deep in your chest. This takes about 30 minutes. You will be given a pretreatment with a bronchodilator medication, and then inhale the mist for at least 1, and up to 3, 7 minute periods. Then you are asked to cough up some sputum from your chest, into a sample cup. Inhalation of the mist can cause coughing and sore throat but pretreatment with the bronchodilator should minimize these side effects. Spirometry is repeated after each inhalation of mist to detect any change in your airway size, or bronchoconstriction. If bronchoconstriction occurs, you will immediately be given a bronchodilator to reverse it. The sputum will be analyzed for markers of inflammation characteristic of your asthma.

At those same visits you will also have approximately 25 mL (2 tablespoons) of blood taken which will be analyzed for markers of inflammation called cytokines. You will also answer a questionnaire to determine how asthma and allergies affect your daily living. You will undergo a physical exam and receive education on how to control your asthma and how to properly use your inhalers.

At the beginning of the study and at the end of the study we will ask that you come in for another visit to do a methacholine challenge breathing test. The challenge involves you breathing a mist that contains a bronchoconstrictor (methacholine) and then performing spirometry to measure the flow and volume of air in your lungs. You will breathe several different mists, of increasing concentrations of the bronchoconstrictor, until a change in your flow measurement is found. This test measures how sensitive your airways are and takes about 1 hour. You may feel some tightness in your chest and/or some wheezing as a result of the challenge, but you will be given bronchodilator medication to reverse the effects of the bronchoconstrictor. You will be closely monitored with spirometry to ensure your safety during this test.

Risks The potential side effects of CLA are minimal. In previous human studies the main complaint was that of gastrointestinal disturbances; mainly bloating and increased gas. 12% of people receiving CLA complained of gastrointestinal disturbances, compared to 6% of people receiving olive oil placebo.

If you are a female of childbearing potential and are pregnant or nursing you cannot be involved in this study, as the effects of CLA on the embryo and fetus are not known. If you become pregnant during the study you must inform the study personnel immediately and your study treatment will be discontinued.

Confidentiality All of the data collected regarding you will be kept in a secure database in the McDonald Research Wing, where it can be accessed by authorized individuals only for this study. No personal information such as your name or address will be included in the database; you will be identified by a code number only.

These investigations are for research only; no individual results will be returned to you or your doctor. Participation in this study is completely voluntary. You may refuse to participate, or you may withdraw from the study at any time without prejudice to your medical treatment.

Benefit There may be no direct benefit to you in participating in this study, but you will be helping us advance our knowledge of lung disease for the benefit of future patients.

Compensation You will be compensated for your time and effort by payment of $25 for your screening visit and $50 for each set of study visits (sputum induction and breathing tests).

ELIGIBILITY:
Inclusion Criteria:

Mild asthma - FEV1 > 70% predicted Positive methacholine challenge

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2002-05; Primary Completion 2002-05 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
PC20 - methacholine sensitivity | 12 weeks

SECONDARY OUTCOMES:
Quality of life (QoL), body mass index (BMI), systemic cytokine levels, and adverse events. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Delbert Dorscheid, MD, Ph.D, Principal Investigator — University of British Columbia; Ruth MacRedmond, MD, FRCPC, Study Director — University of British Columbia
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada